CLINICAL TRIAL: NCT03604250
Title: The January Application NUtritional Study: Health Optimization by Wearable Devices - a Pilot Trial
Brief Title: The January Application NUtritional Study (JANUS)
Acronym: JANUS
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study protocol under revision.
Sponsor: January, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-44
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: This is a pilot trial with a single group of 14 participants: 10 with prediabetes or at least 2 of the metabolic syndrome criteria (half males, half females) 4 healthy people (do not have prediabetes nor any of the metabolic syndrome criteria) of 11 weeks (77 days) duration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle plus prebiotics (Experimental): Research participants will be asked to wear health monitoring devices, including a continuous glucose monitoring device and an Apple watch. They may be prompted to perform lifestyle modifications aimed at better understanding their health parameters, based on the results obtained from the wearable devices and other tests. During the last 3 weeks of the study, research participants may be asked to take a personalized prebiotic supplement, up to once/day.
  Interventions: Dietary Supplement: Lifestyle plus prebiotic supplement

INTERVENTIONS:
Dietary Supplement: Lifestyle plus prebiotic supplement — Research participants will be asked to wear health monitoring devices, including a continuous glucose and heart-rate monitors. They may be prompted to perform lifestyle modifications aimed at better understanding their health parameters, based on the results obtained from the wearable devices and other tests. During the last 3 weeks of the study, research participants may be asked to take a personalized prebiotic supplement, up to once/day.

SUMMARY:
Human beings react differently to changes in diet, exercise, and sleep patterns. The goal of this study is to (1) learn how individuals react to lifestyle choices and suggestions by examining a small group of people with similar health and lifestyle profiles; and (2) to develop algorithmic policies (male/female) that will help people optimize their health through lifestyle interventions and supplementation with prebiotics.

DETAILED DESCRIPTION:
Human beings react differently to changes in diet, exercise, and sleep patterns. The goal of this study is two-fold and consists of two phases involving the same subjects. In the first phase, the study aims to learn how individuals react to lifestyle choices and suggestions by examining a small group of people with similar health and lifestyle profiles. Specifically, how their food choices, physical activity pattern, sleep pattern, and stress levels affect glucose metabolism, stress response, inflammation, and microbiome composition.

In the second phase of the study, the investigator's goal is to use the data collected to develop algorithmic policies that will help people optimize their health through lifestyle interventions and supplementation with prebiotics. The ultimate goal is to achieve optimization of glucose and stress regulation, inflammation state, and microbiome composition by observing real-time variations of these regulatory systems through the use of wearable health-monitoring devices and providing lifestyle suggestions via a mobile application.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Both women and men
* Age: between 30 and 60 years
* Ethnicity and race: All
* Are prediabetic (HbA1c </= 6.4 in the past 3 months), or have a fasting plasma glucose > 110 mg/dL, or have 2 of the metabolic syndrome criteria as defined by the International Diabetes Federation (IDF):

Central obesity, defined as waist circumference >/ = 94 cm for men and >/= 80 cm for women, or a BMI > 30 kg/m2 plus any two of the following four factors:

* Raised triglycerides: >/= 150 mg/dL or specific treatment for this lipid abnormality
* Reduced HDL cholesterol:
* Men: < 40 mg/dL
* Women: < 50 mg/dL
* Raised blood pressure (BP): systolic BP >/= 130 mmHg or diastolic BP >/= 85 mmHg, or treatment of previously diagnosed hypertension
* Raised fasting plasma glucose (FPG): FPG >/= 100 mg/dL

  * Have elevated levels of at least one of the following inflammatory markers: C-Reactive Protein (CRP), Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF), Interferon gamma (IFN-G), Interleukins (IL-1b, IL-2, IL-6, IL-8, IL-10, IL-12p70), and Tumor necrosis factor alpha (TNF-a).
  * Are able to utilize a smart-phone and own an Android (v18+) or Apple phone (i0S9+)
  * Are willing to being tracked, provide multiple samples and wear a glucose monitor and a smartwatch 24 hours/day for 77 days
  * Are willing to perform finger-stick blood draws
  * Are willing to limit swimming to a maximum of 30 minutes per session during the trial
  * Are willing to limit traveling to the weekend days
  * Live in the vicinity of January Inc office and/or MBC Biolabs (Approximately 25 mile radius)
  * Are available for two, 2-4-hour meetings (study orientation and study close-out)
  * Eat a steady, consistent diet on a daily basis (see dietary exclusions below)
  * Are able to run for the time required to establish VO2 max (3-20 minutes).
  * Have the ability and willingness to give written informed consent

Exclusion Criteria:

* Smokers
* BMI =/> 40
* Actively losing weight
* Unstable diet (defined as having made any major changes to usual diet such as eliminating or significantly increasing a major food group)
* Use of the following medications:

  * Blood thinners (i.e. warfarin/Coumadin, clopidogrel/Plavix)
  * Daily oral corticosteroids
  * Hypoglycemic medication (i.e. Precose, Metformin, Avandia, Victoza)
  * Weight loss medication
  * Digoxin/Lanoxin
  * Lithium/Lithobid
  * Theophylline/Theo 24
* Use of the following supplements, unless they agree to discontinue starting 30 days prior to the trial: any nutritional supplements containing antioxidants (examples: multi-vitamins, antioxidant combinations, or any supplement containing vitamin C, vitamin E, beta-carotene or other carotenoids, or selenium), and fish oil/cod liver oil, flaxseed oil, and supplements containing Conjugated linoleic acid (CLA)/Gamma-linolenic acid (GLA) or turmeric.
* Use of antibiotics, antifungals/antiparasitics in the last 30 days
* Use of probiotic or prebiotic supplements in the last 30 days
* People allergic to: adhesives and/or prebiotics used in the trial
* Pregnant, lactating, have given birth in the past 6 months, or are planning to get pregnant in the next 4 months
* Self-reported health conditions:

  * Diabetes (T1D or T2D)
  * Inflammatory Bowel Disease (Crohn's, Ulcerative Colitis)
  * Gastroenteritis, colitis or gastritis
  * Active, uncontrolled Clostridium difficile infection or H. pylori (untreated)
  * Recent heart attack (past 6 months), history of arrhythmias or cerebrovascular disease
  * Undergoing treatment for, or underwent treatment for cancer in the past 6 months
  * Esophageal, stomach colon or pancreatic cancer
  * Liver disease, other than fatty liver disease
  * Immunosuppression or immunodeficiency
  * Positive test for HIV, Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV)
  * Musculoskeletal disorder that would preclude you from performing moderate physical activity
  * LDL cholesterol =/> 190 mg/dL
  * Triglycerides (TG) =/> 450 mg/dL
  * Adrenalectomy
  * Pituitary tumor
  * Hypothalamic disease
  * Stage 3 kidney disease or worse
  * Celiac disease confirmed by blood test or biopsy
  * Insulinoma
  * Cushing's disease
  * Hyperthyroidism
  * Acromegaly
  * Pheochromocytoma
  * Addison's disease
  * Galactosemia
  * Glycogen storage disease
  * Hereditary fructose intolerance
  * Psychotic disorders or bipolar disorders
  * Current eating disorder
* History of bariatric surgery, gallbladder removal, small bowel resection, or extensive bowel resection
* Hospitalization for depression in past 6 months
* Self-reported alcohol or substance abuse within the past 12 months
* Current consumption of more than 14 alcoholic drinks per week, and/or current acute treatment or rehabilitation program for these problems
* Self-reported inability to walk two blocks
* Restrictive diets (i.e. vegetarians, vegans, or very restrictive diets, i.e. Paleo, Atkins, Ornish or ketogenic diets)
* Planned travel (outside of weekends) over the course of the study (77 days) (weekend travel is ok)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Total Health Score (THS) | 11 weeks
  The primary outcome of the study is the calculation of a Total Health Score (THS) which will include scores of body composition, glucose and stress regulation, inflammation state, and microbiome composition, based on the following data:
  * Anthropometrics
  * Blood pressure
  * Heart Rate
  * Glucose
  * Hemoglobin A1c
  * Metabolic panel
  * Complete Blood Count
  * Glomerular Filtration Rate
  * Inflammatory markers
  * Serum lipids
  * Thyroid-stimulating hormone
  * Blood ketones
  * Cortisol
  * C-peptides
  * Metagenomics
  * Metabolomics
  * 16S rRNA sequencing
  * Human genome assays (SNP, Exome+)

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Perelman, MS, RD, CDE, Principal Investigator — January, Inc.
Locations (1):
- January, Inc., Menlo Park, California, United States

IPD SHARING:
Plan to Share IPD: No